CLINICAL TRIAL: NCT03285243
Title: Effect of Monochromatic Light on Incidence of Emergence Delirium in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Adam Adler MD, MS, FAAP, Assistant Professor of Anesthesiology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-39878
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Results first posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Emergence Delirium; Anesthesia Emergence Delirium
Keywords: Delirium, anesthesia, pediatrics
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Intervention Model Description: This is a double blinded randomized control trial. The placebo arm will serve as the control group. After enrollment and consent, each patient will be randomized to either placebo or intervention group. 110 sealed envelopes randomizing patients to the exposure group A (monochromatic light) or bulb B (placebo) white light bulb with blue outer coating.
Who Masked: Participant, Care Provider
Masking Description: After enrollment and consent, each patient will be randomized to either placebo or intervention group. 110 sealed envelopes randomizing patients to the exposure group A (monochromatic light) or bulb B (placebo) white light bulb with blue outer coating. The recover room nursing staff will evaluate the patient using the PAED standard emergence delirium scale unaware of which light is monochromatic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Blue light - non monochromatic (Sham Comparator)
  Interventions: Device: Monochromatic blue light
- Monochromatic blue light (Experimental)
  Interventions: Device: Monochromatic blue light

INTERVENTIONS:
Device: Monochromatic blue light — Exposure to monochromatic light for the first 30 minutes in the recovery period after anesthesia to assess incidence of emergence delirium as noted by the PAED scale

SUMMARY:
Emergence delirium/emergence agitation (ED/EA) is a behavioral phenomenon of unclear etiology consisting of short lived behavioral changes that can be both traumatic to families and pose a safety risk to patients and staff. ED is characterized by a variety of presentations, including crying, excitation and agitation, that occur during the early stage of recovery from general anesthesia, generally in the first 30 minutes. Emergence delirium occurs in children of all ages following an anesthetic with halogenated agents (e.g. sevoflurane/isoflurane) with or without having undergone a surgical procedure (e.g. MRI patients). Presently, the treatment for ED is to revert the patient back to a hypnotic state mainly with sedatives so that they may "reset" themselves postulating that by re-inducing a hypnotic state, the brain has time to resolve this issue. The hypothesis of this study is that during ED, there is failure of organized EEG activity, especially alpha wave activity and that by enhancing alpha activity, the incidence of ED may be reduced without the need for additional pharmaceuticals which may be costly, delay recovery and are not without adverse effects specifically cardiopulmonary depression through the use of blue monochromatic light.

DETAILED DESCRIPTION:
Emergence delirium/emergence agitation (ED/EA) is a behavioral phenomenon of unclear etiology consisting of short lived behavioral changes that can be both traumatic to families and pose a safety risk to patients and staff. ED is characterized by a variety of presentations, including crying, excitation and agitation, that occur during the early stage of recovery from general anesthesia, generally in the first 30 minutes. Involuntary activity in the bed and even thrashing about during an episode of ED can lead to dislodgement of IV cannulas, surgical dressings and or surgically placed items such as drains and catheters. Emergence delirium occurs in children of all ages following an anesthetic with halogenated agents (e.g. sevoflurane/isoflurane) with or without having undergone a surgical procedure (e.g. MRI patients). Electroencephalograms (EEG) in patients experiencing emergence delirium show diffuse background slowing. Presently, the treatment for ED is to revert the patient back to a hypnotic state mainly with sedatives so that they may "reset" themselves postulating that by re-inducing a hypnotic state, the brain has time to resolve this issue. The hypothesis of this study is that during ED, there is failure of organized EEG activity, especially alpha wave activity and that by enhancing alpha activity, the incidence of ED may be reduced without the need for additional pharmaceuticals which may be costly, delay recovery and are not without adverse effects specifically cardiopulmonary depression.

Monochromatic light (ML) has been used in a variety of clinical and non-clinical applications to affect a variety of changes. Exposure to light of short wavelength within the visible spectrum (450-470nm) has been associated with effects on circadian rhythm, neuroendocrine and neurobehavioral changes and enhanced cognitive performance. Blue ML has been studied safely to enhance work-place alertness and productivity. Clinically, blue ML has been used safely for decades in the neonatal intensive care unit to treat jaundice.

Blue ML, has been known to suppress melatonin secretion and enhance alertness and workplace performance. The effect occurs within the retinal photoreceptive ganglion cells which mediate the observed responses. The effect is even present in visually blind persons lacking outer retinal function. Short exposure to bursts of blue light has revealed enhanced neural activity on functional MRI. Use of blue ML has been shown to enhance EEG activity in the alpha range (awake range) compared with light of greater wavelengths. Using blue ML in the operating room may enhance alpha EEG activity, (a circadian marker for alertness) it may be possible to reduce the incidence of emergence delirium in the post-operative period and therefore the amount of (non-pain) sedative medication needed in recovery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist Classification of 1,2
* Patients ages 2-6 years
* Routine tonsillectomy and adenoidectomy

Exclusion Criteria:

American Society of Anesthesiology classification other than 1,2; history of migraine headaches; ocular disorders; seizure history; psychiatric conditions; anxiety; parental refusal; developmental delay; patients on medication for attention deficit disorders or caffeine stimulants; Patients with contraindications to receiving inhalation agents; Use of premedication with midazolam or dexmedetomidine;

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Adler, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas childrens Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Patient Data will be kept on file and disclosed at discretion of the PI in accordance with Baylor College of Medicine regulations

REFERENCES:
- [Derived] Adler AC, Nathanson BH, Chandrakantan A. Monochromic light reduces emergence delirium in children undergoing adenotonsillectomy; a double-blind randomized observational study. BMC Anesthesiol. 2021 Sep 8;21(1):217. doi: 10.1186/s12871-021-01435-1. PMID 34496743

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was performed between November 3, 2017 and June 2, 2020
Period: Overall Study
Arm/Group | Blue Light - Non Monochromatic | Monochromatic Blue Light
Started | 52 | 52
Completed (found to have met exclusion criteria after enrollment) | 52 | 51
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blue Light - Non Monochromatic | Monochromatic Blue Light | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 52 | 52 | 104
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.2 (1.4) | 4.7 (1.3) | 4.5 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 28 | 28 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 52 | 52 | 104
Region of Enrollment [Number; unit: participants]
  United States | 52 | 52 | 104

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Emergence Delirium Following Anesthesia in Children
Description: Assessment if monochromatic light reduces the absolute incidence of emergence delirium following general anesthesia (as a binary: emergence delirium vs. no emergence delirium)
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Blue Light - Non Monochromatic | Monochromatic Blue Light
Number analyzed (Participants) | 52 | 52
Participants | 17 | 3
Statistical Analysis 1: Comparison: Blue Light - Non Monochromatic vs Monochromatic Blue Light; Test type: Other; p = 0.001, Chi-squared — A priori, All p-values < 0.05 were considered statistically significant

2. Secondary Outcome: Number of Participants With PAED Scale Score of 12 or More for 30 Minutes After Baseline
Description: Assessment of Pediatric Emergence Delirium Scale (PAED) scale scores at varying points during the initial recovery phase in patients exposure to monochromatic light vs. sham Pediatric Emergence Delirium Scale scored ranges from a Minimum of 2 to a maximum of 20. Higher scores are associate with emergence delirium and agitation indicating a worse outcome
Time Frame: 30 minutes
Population: Patient had Emergence Delirium or a PAED Scale Score of 12 or more for 30 minutes after Baseline(n, %)
Measure: Count of Participants; unit: Participants
Arm/Group | Blue Light - Non Monochromatic | Monochromatic Blue Light
Number analyzed (Participants) | 52 | 52
Participants | 27 | 12
Statistical Analysis 1: Comparison: Blue Light - Non Monochromatic vs Monochromatic Blue Light; Test type: Other; p = 0.002, Regression, Logistic — a priori, all p-values < 0.05 were considered statistically significant

ADVERSE EVENTS:
Time Frame: 1 hour
Description: The definitions of adverse events does not differ from clinical trials.gov definitions
Arm/Group | Blue Light - Non Monochromatic | Monochromatic Blue Light
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/43/NCT03285243/Prot_SAP_003.pdf